CLINICAL TRIAL: NCT00389727
Title: A Dose Escalation Study With Intensity Modulated Radiation Therapy (IMRT) in Moderately Advanced (T2N0, T2N1, T3N0) Squamous Cell Carcinomas (SCC) of the Oropharynx, Larynx and Hypopharynx Using a Simultaneous Integrated Boost (SIB) Approach.
Brief Title: Simultaneous Integrated Boost (SIB)- IMRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-01avr-074
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Patients (Experimental): Radiotherapy Patients
  Interventions: Drug: Radiotherapy
- Group 2 (No Intervention)

INTERVENTIONS:
Drug: Radiotherapy — Radiotherapy
  Arms: Group 1 Patients

SUMMARY:
The objective of the study is to assess the feasibility of increasing dose of irradiation with IMRT using a SIB approach over 6 weeks.

The primary endpoint of the study will be acute toxicity assessed during treatment and during the first 3 months following the completion of radiotherapy The secondary endpoint will include loco-regional control, disease-free survival, survival and late toxicity at 2 years after completion of radiotherapy

DETAILED DESCRIPTION:
Loco-regional failures remain a major concern following irradiation of locally advanced head and neck cancers. This has led radiation oncologists to investigate novel approaches offering better therapeutic indexes. Modification of dose fractionation schedules can improve the therapeutic outcome by using accelerated or hyperfractionated regimes -Ang, 1990; Ang, 1998; Fu, 2000; Gwozdz, 1997-. Intensity Modulated Radiation Therapy (IMRT) technique allows the planning and irradiation of different targets at different dose levels in a single treatment session, instead of successive treatment plans. With conventional 2D radiotherapy, both normal tissues and tumors are irradiated with a similar dose per fraction of 1.8-2 Gy, whereas with IMRT dose gradients are introduced in such a manner that normal tissues receive a much lower dose per fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with squamous cell carcinoma of the oropharynx, hypopharynx and larynx
* Stage T2-N0-M0, T2-N1-M0 or T3-N0-M0
* World Health Organization (WHO) Performance Status of 0 or 1 or Karnofsky performance status ≥ 70.
* Provision of written informed consent

Exclusion Criteria:

* Second primary tumor at the time of diagnosis
* Previous history of malignant tumor in the last five years except basal cell carcinoma and carcinoma in situ of the cervix
* Previous treatment with surgery, radiotherapy or chemotherapy for head and neck malignancy
* Any evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease), or psychological disorder
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-09-24 (Actual); Primary Completion 2008-05-26 (Actual); Study Completion 2008-05-26 (Actual)

PRIMARY OUTCOMES:
acute toxicity | during treatment and during the first 3 months following the completion of radiotherapy
  acute toxicity

SECONDARY OUTCOMES:
composite endpoint | from ratiotherapy until 2 years after completion of radiotherapy
  composite including loco-regional control, disease-free survival, survival and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gregoire, MD, PhD, Study Chair — Cliniques universitaires Saint Luc Brussels Belgium; Philippe Maingon, MD, PhD, Study Chair — Centre George-François Leclerc Dijon, France; Sandra Nuyts, MD, Principal Investigator — University hospital Gasthuisberg, Katholiek universiteit van Leuven; Gilles Calais, MD, PhD, Principal Investigator — CHU de Tours, Bretonneau; Antoine Serre, MD, Principal Investigator — centre Val d'Aurelle, Montpellier
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium